CLINICAL TRIAL: NCT01191125
Title: Evaluation of an Oral Nutritional Supplement Containing AN777 in Malnourished and Frail Subjects
Brief Title: Evaluation of an Oral Nutritional Supplement Containing AN777
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BK94
Record Dates: First submitted 2010-08-27; First posted 2010-08-30 (Estimated); Last update posted 2013-03-07 (Estimated); Status verified 2013-03

CONDITIONS: Malnutrition; Sarcopenia
MeSH Terms: conditions — Malnutrition; Sarcopenia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- medical food with AN777 (Experimental)
  Interventions: Other: medical food with AN777
- oral nutritional formula (Active Comparator)
  Interventions: Other: oral nutritional formula

INTERVENTIONS:
Other: medical food with AN777 — Two(220 mL)servings every day for six months
  Arms: medical food with AN777
Other: oral nutritional formula — Two (220 mL) servings daily for six months
  Arms: oral nutritional formula

SUMMARY:
To evaluate the effect of an experimental oral nutritional supplement containing AN777 compared to another oral nutritional supplement in a malnourished, elderly population.

ELIGIBILITY:
Inclusion Criteria:

Subject (male or female) is > or equal to 65 and < or equal to 90 years of age

Subject is ambulatory

Subject has a Subjective Global Assessment of B or C

Subject has gait speed <0.8 m/s AND/OR low hand-grip strength

Subject has Class 1 or Class 2 sarcopenia

Subject agrees to refrain from starting a resistance exercise program

Exclusion Criteria:

Subject has type 1 or type 2 diabetes

Subject has inflammatory disease with elevated high sensitivity C-reactive protein

Subject has renal function impairment

Subject reports gastrointestinal disorder (severe chronic diarrhea, nausea, vomiting) that would preclude ingestion of the study product; an obstruction of the gastrointestinal tract, inflammatory bowel disease; short bowel syndrome or other major gastrointestinal disease

Subject reports of current active malignant disease or other significant medical diagnoses.

Subject reports a history of allergy to any of the ingredients in the study products

Subject reports currently taking medications/dietary supplements/substances that could profoundly modulate metabolism or weight.

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 331 (Actual)
Dates: Start 2011-02; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Knee extensor strength | Six months

SECONDARY OUTCOMES:
Leg muscle mass | Six months
Body Weight | Six months
Functional measures | Six months

CONTACTS AND LOCATIONS:
Overall Officials: Vikkie Mustad, PhD, Study Chair — Abbott Nutrition
Locations (23):
- United States (8):
  - University of Alabama, Brimingham, Birmington, Alabama
  - Radiant Research, Inc, Santa Rosa, California
  - Provident Clinical Research, Addison, Illinois
  - Radiant Research, Inc, Chicago, Illinois
  - Radiant Research, Inc., Overland Park, Kansas
  - Creighton University, Omaha, Nebraska
  - Radiant Research, Inc, Cincinnati, Ohio
  - Radiant Research, Inc., Dallas, Texas
- ZNA St. Elisabeth, Antwerp, Belgium
- Italy (2):
  - Catholic University of Rome, Rome
  - University of Verona, Verona
- Althian - Research Management Center, Monterrey, Nuevo León, Mexico
- Poland (4):
  - NSZOZ Unica CR, Dąbrówka
  - Mazowieckie Centrum Badan Klinicznych S.C.., Grodzisk Mazowiecki
  - Tomasz Dabrowski Slaskie Centrum, Katowice
  - Centrum Medyczne Osteomed, Warsaw
- Spain (4):
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Insituto Provincial de Rehabilitacion, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
- University Hospitals, WHO, Geneva, Switzerland
- United Kingdom (2):
  - Imperial College Healthcare NHS Trust, Charing Cross, London
  - University of Nottingham Medical School,, Nottingham

REFERENCES:
- [Derived] Cramer JT, Cruz-Jentoft AJ, Landi F, Hickson M, Zamboni M, Pereira SL, Hustead DS, Mustad VA. Impacts of High-Protein Oral Nutritional Supplements Among Malnourished Men and Women with Sarcopenia: A Multicenter, Randomized, Double-Blinded, Controlled Trial. J Am Med Dir Assoc. 2016 Nov 1;17(11):1044-1055. doi: 10.1016/j.jamda.2016.08.009. PMID 27780567
- [Derived] Hickson M. Nutritional interventions in sarcopenia: a critical review. Proc Nutr Soc. 2015 Nov;74(4):378-86. doi: 10.1017/S0029665115002049. Epub 2015 Apr 29. PMID 25923603